CLINICAL TRIAL: NCT00661739
Title: A Multicentre Phase I-II Study to Investigate the Combination of Bendamustine With Weekly Paclitaxel as First or Second Line Therapy in Patients With Metastatic Breast Cancer
Acronym: RiTa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBG 38
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Metastatic Breast Cancer
Keywords: palliative; Breast cancer; metastatic; Bendamustine; phase I
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Singular Arm (Experimental): Bendamustine treatment
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — Dose-level Bendamustine(mg/m²): I:50; II:60; III:60; IV:70; V:70 Dose-level Paclitaxel (mg/m²): I:60; II:60; III:80; IV:80; V:90 Treatment will be given on day 1,8,15 and repeated on day 29. When the recommended dose has been determined a total of 48 pts will be treated at this dose level.
  Other Names: Ribomustine

SUMMARY:
The aim of the study is to establish a feasible combination of bendamustine and paclitaxel in a weekly schedule. The two agents have different toxicity profiles and are well tolerated when given in a weekly fashion. The combination might be of special interest for elderly patients with hormone insensitive breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures;
* Pathological confirmed primary carcinoma of the breast.
* Locally advanced or metastatic disease
* Up to one previous palliative chemotherapy that did not contain docetaxel or paclitaxel. Previous adjuvant treatment with taxanes is allowed when the last application of the taxane was given at least 1 year before entering the trial.
* Patients must have either measurable or non-measurable lesions according to the WHO criteria
* At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiated field or there must be pathological proof of progressive disease.
* Complete radiological and clinical tumor assessment within 4 weeks prior to registration performed as clinically indicated
* Karnofsky-Index ≥ 60 %
* Age ≥ 18 years
* Absolute neutrophil count ≥ 1,500 cells/µl, platelets ≥ 100,000/µl, and hemoglobin ≥ 9 g/dl
* Bilirubin within normal limits; evaluation of transaminases and alkaline phosphatase ≤ 5x upper normal limit
* Serum creatinine ≤ 2.0 mg/dl
* Normal left ventricular ejection fraction (LVEF) by echocardiogramme
* Patients of childbearing potential, pregnancy test must be negative
* If fertile effective contraception must be used throughout the study

Exclusion Criteria:

* Known or suspected hypersensitivity reaction to the investigational compounds or incorporated substances;
* Concurrent immunotherapy or hormonal treatment for cancer (Bisphosphonates may be continued)
* Symptomatic parenchymal brain metastases not responding to treatment
* Life expectancy less than 3 months
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study
* Concurrent treatment with other experimental drugs or any other anti-cancer therapy within the last 28 days;
* History of congestive heart failure or other significant uncontrolled cardiac disease
* Pregnant or nursing women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-07; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The phase I part of the trial should evaluate the maximal tolerated dose (MTD) for the combination of bendamustine with paclitaxel. | end of cycle 2 of the 6th patient of the assumed highest dose level

SECONDARY OUTCOMES:
To determine the objective response rate (phase II part) | EOT last patient (phase II part)